CLINICAL TRIAL: NCT00593970
Title: Knowledge Possessed by Pregnant Women Regarding Influenza Vaccination During Pregnancy
Brief Title: Influenza Vaccine in Pregnancy Part 2
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 06-190 part2
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Influenza; Pregnancy
Keywords: influenza; vaccine; pregnancy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All women presenting to our prenatal clinic and postpartum floor during the study period.

SUMMARY:
Pregnant women have limited knowledge regarding influenza, its implications during pregnancy, and recommendations for vaccination during pregnancy. The researchers plan to distribute an information pamphlet to women in a prenatal clinic, offer the vaccine during prenatal visits, and then give a questionnaire on the postpartum floor assessing knowledge.

The researchers hypothesize that with education intervention, knowledge scores on the questionnaire will be higher than those from last year, when no education was provided.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women

Exclusion Criteria:

* known hypersensitivity to influenza vaccine

Ages: 14 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A multi-ethnic group of pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Knowledge scores on our questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Yudin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada